CLINICAL TRIAL: NCT06595186
Title: A Multicenter, Single Arm, Open-label, Dose-escalation Phase 2 Study of JK-1201I Combined with Adjuvant Temozolomide in Patients with Newly Diagnosed Glioblastoma Multiforme (GBM) After Surgery and Concomitant Radio-chemotherapy
Brief Title: JK-1201I Combined with Adjuvant Temozolomide in Patients with Newly Diagnosed Glioblastoma Multiforme (GBM)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: JenKem Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JK-1201I-202
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Glioblastoma Multiforme (GBM)
Keywords: glioblastoma multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation Cohort (Experimental): Participants will receive JK-1201I as an intravenous (IV) infusion at each 14-day cycle (Q2W) until a treatment discontinuation criterion is met as specified in the protocol. Escalating doses of JK-1201I will be evaluated by the traditional 3+3 design.
  Temozolomide will be administered per drug label.
  Interventions: Drug: JK-1201I; Drug: Temozolomide (TMZ)
- Dose Expansion Cohort (Experimental): Participants will receive JK-1201I as an intravenous (IV) infusion as the recommended Phase 2 dose at each 14-day cycle (Q2W) until a treatment discontinuation criterion is met as specified in the protocol.
  Temozolomide will be administered per drug label.
  Interventions: Drug: JK-1201I; Drug: Temozolomide (TMZ)

INTERVENTIONS:
Drug: JK-1201I — JK-1201I will be administered.
Drug: Temozolomide (TMZ) — Temozolomide will be administered.

SUMMARY:
This study was designed to evaluate the safety, tolerability, efficacy and pharmacokinetics of JK-1201I combined with adjuvant temozolomide in patients with newly diagnosed glioblastoma multiforme after surgery and concomitant radio-chemotherapy.

DETAILED DESCRIPTION:
This is a multicenter, single arm, open-label, dose-escalation phase 2 study of JK-1201I combined with adjuvant temozolomide in patients with newly diagnosed glioblastoma multiforme (GBM) after surgery and concomitant radio-chemotherapy Patients will receive JK-1201I combined with temozolomide until disease progression.

The primary objective of this study is to assess the safety of JK-1201I combined with adjuvant temozolomide in patients with newly diagnosed glioblastoma multiforme after surgery and concomitant radio-chemotherapy.

The secondary objectives of the study are to further evaluate the efficacy and pharmacokinetic profiles of JK-1201I.

ELIGIBILITY:
Inclusion

Participants must meet all the following criteria to be eligible for randomization into the study:

1. Male or female aged ≥18 years and ≤75 years.
2. Patients newly diagnosed with glioblastoma either by imaging or pathology testing, Gross total resection equal to or greater than 80%.
3. Patients must finish concurrent chemo-radiotherapy (CCRT) no sooner than 4 weeks and no later than 6 weeks.
4. Stable dose or reduced dose of corticosteroid for more than 2 weeks.
5. Karnofsky score ≥ 70.
6. Life expectancy > 12 weeks.
7. Adequate biological function.
8. Men or women should be using adequate contraceptive measures during the study and for 6 months following the last dose of investigational product.
9. Sign and date the informed consent form prior to the start of any study-specific qualification procedures.
10. MGMT unmethylation (only for Dose Expansion Cohort).

Exclusion

Participants who meet any of the following criteria will be disqualified from entering the study:

1. Patients who received anti-tumor therapy except for concurrent chemo-radiotherapy (CCRT).
2. Patient diagnosed with brain stem and spinal cord tumor as the primary tumor.
3. Hypersensitivity to any ingredient of JK-1201I.
4. Severe, uncontrolled or active cardiovascular diseases within the past 6 months.
5. Inability to take medication by oral or presence of clinically significant gastrointestinal abnormalities that may affect absorption of investigational product.
6. Uncontrolled seizures.
7. Patient receiving prohibited medications and that cannot be discontinued at least 2 weeks prior to the start of treatment.
8. Severe or uncontrolled high blood pressure.
9. Unresolved toxicity from prior anti-tumor therapy.
10. Women who are pregnant or Breast-feeding. 11 Positive human immunodeficiency virus antibody, active hepatitis B virus infection, or active hepatitis C virus infection.

12. Have participated in another clinical trial within 4 weeks prior to informed consent form.

13. History of mental disorders. 14. Other conditions that the investigator considers unsuitable to participate in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2026-08-16 (Estimated); Study Completion 2026-12-16 (Estimated)

PRIMARY OUTCOMES:
Incidence and Grade of Participants with Adverse Events or Serious Adverse Events | From the date of first dose to the end of safety follow-up; Up to 12 months.
  Adverse Events (AEs) or Serious Adverse Events (SAEs) are assessed based on NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) Assessed by Investigators | From the date of randomization to documented progressive disease, death, lost to follow-up, or withdrawal by the participant; Up to 12 months.
  Progression-free Survival (PFS) is defined as the time interval from the randomization to disease progression or death due to any cause.
Overall survival (OS) | From the date of randomization to the date of death due to any cause; Up to 12 months.
  Overall survival (OS) is defined as the time interval from randomization to death due to any cause.
Pharmacokinetic Parameter Area Under the Plasma Concentration-Time Curve for JK-1201I, Irinotecan, SN38 and SN38G | Up to 6 months.
  Area under the plasma concentration-time curve up to the last quantifiable time point (AUClast) and area under the plasma concentration-time curve dosing interval (AUCtau) will be assessed using Non-linear mixed effect modeling.
Pharmacokinetic Parameter Maximum Concentration for JK-1201I, Irinotecan, SN38 and SN38G | Up to 6 months.
  Maximum concentration (Cmax) will be assessed using Non-linear mixed effect modeling.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, China